CLINICAL TRIAL: NCT00564902
Title: Randomized, Double Blind, Lutein Controlled Study of Zeaxanthin and Visual Function in Atrophic Age Related Macular Degeneration Patients
Brief Title: The Zeaxanthin and Visual Function Study
Acronym: ZVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chrysantis, Inc. (Industry)
Collaborators: Kowa Company, Ltd. (Industry); IMAGE TECHNOLOGIES INC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CHRY1; IRB 07-046 (Other: Edward Hines Jr. VA Hospital/North Chicago VAMC)
Record Dates: First submitted 2007-11-27; First posted 2007-11-29 (Estimated); Results first posted 2012-03-29 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Age Related Macular Degeneration; Cognition Disorders
Keywords: Macular Pigment Optical Density; Skin Carotenoids; Lipofuscin; Photostress (Glare Recovery); Visual Field Progression; Contrast Sensitivity; Color Vision; Cognitive Function
MeSH Terms: conditions — Macular Degeneration; Cognition Disorders | interventions — Zeaxanthins; Lutein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lutein (Placebo Comparator): 9 mg of Lutein for 12 months
  Interventions: Dietary Supplement: Lutein
- Zeaxanthin and Lutein (Active Comparator): 3R 3'R Zeaxanthin 8 mg, Lutein 8 mg per day during 12 months
  Interventions: Dietary Supplement: Lutein and Zeaxanthin
- Zeaxanthin (Active Comparator): 3R 3'R Zeaxanthin 8 mg per day during 12 months
  Interventions: Drug: 3R 3'R Zeaxanthin

INTERVENTIONS:
Drug: 3R 3'R Zeaxanthin — 8 mg per day during 12 months
  Other Names: EZEyes
  Arms: Zeaxanthin
Dietary Supplement: Lutein — 9 mg of Lutein during 12 months
  Arms: Lutein
Dietary Supplement: Lutein and Zeaxanthin — 8 mg of lutein and 8 mg of Zeaxanthin administered during 12 months
  Arms: Zeaxanthin and Lutein

SUMMARY:
To evaluate if supplementation of zeaxanthin (with or without Lutein) is beneficial to patients with early and moderate Atrophic Age Related Macular Degeneration.

DETAILED DESCRIPTION:
To evaluate whether or not zeaxanthin supplementation raises macular pigment optical density (MPOD). Previous research has shown MPOD to mirror visual benefits for patients with age related atrophic macular degeneration (AMD) having visual symptoms (decreased visual acuity, contrast sensitivity, photostress glare recovery and National Eye Institute Visual Function Questionnaire 25 scores), but lower risk National Eye Institute (NEI) / Age Related Eye Disease Study (AREDS) characteristics.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of atrophic AMD (ICD9 362.51) by stereo bio-ophthalmoscopy and at least one vision degrading visual-psychophysical abnormality associated with AMD in one or both eyes.
* clear non-lenticular ocular media (cornea, aqueous and vitreous)
* free of advanced glaucoma and diabetes or any other ocular or systemic disease that could affect central or parafoveal macula visual function

Exclusion Criteria:

* high risk retinal characteristics for advanced AMD or advanced AMD for which existing medical / surgical options are available
* presence of ophthalmologically significant active exudative, AMD pathology by fluorescein angiography but also a single large drusen, >15, multiple intermediate drusen, parafoveal geographic atrophy or loss of vision in one eye due to advanced AMD
* recent (within 6 months) cataract or retinal surgery
* taking photosensitizing drugs such as phenothiazines and chloroquine
* having taken lutein or zeaxanthin supplements within the past six months.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-11; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Richer, Ph. D., Principal Investigator — North Chicago VA Medical Center; William Stiles, M.D., Study Director — North Chicago VA Medical Center
Locations (1):
- North Chicago VA Medical Center, North Chicago, Illinois, United States

REFERENCES:
- [Background] Delcourt C, Carriere I, Delage M, Barberger-Gateau P, Schalch W; POLA Study Group. Plasma lutein and zeaxanthin and other carotenoids as modifiable risk factors for age-related maculopathy and cataract: the POLA Study. Invest Ophthalmol Vis Sci. 2006 Jun;47(6):2329-35. doi: 10.1167/iovs.05-1235. PMID 16723441
- [Background] Schalch W, Cohn W, Barker FM, Kopcke W, Mellerio J, Bird AC, Robson AG, Fitzke FF, van Kuijk FJ. Xanthophyll accumulation in the human retina during supplementation with lutein or zeaxanthin - the LUXEA (LUtein Xanthophyll Eye Accumulation) study. Arch Biochem Biophys. 2007 Feb 15;458(2):128-35. doi: 10.1016/j.abb.2006.09.032. Epub 2006 Nov 7. PMID 17084803
- [Background] Richer S, Stiles W, Statkute L, Pulido J, Frankowski J, Rudy D, Pei K, Tsipursky M, Nyland J. Double-masked, placebo-controlled, randomized trial of lutein and antioxidant supplementation in the intervention of atrophic age-related macular degeneration: the Veterans LAST study (Lutein Antioxidant Supplementation Trial). Optometry. 2004 Apr;75(4):216-30. doi: 10.1016/s1529-1839(04)70049-4. PMID 15117055
- [Background] Richer S, Devenport J, Lang JC. LAST II: Differential temporal responses of macular pigment optical density in patients with atrophic age-related macular degeneration to dietary supplementation with xanthophylls. Optometry. 2007 May;78(5):213-9. doi: 10.1016/j.optm.2006.10.019. PMID 17478338
- [Background] Leung IY, Sandstrom MM, Zucker CL, Neuringer M, Max Snodderly D. Nutritional manipulation of primate retinas. IV. Effects of n--3 fatty acids, lutein, and zeaxanthin on S-cones and rods in the foveal region. Exp Eye Res. 2005 Nov;81(5):513-29. doi: 10.1016/j.exer.2005.03.009. PMID 15916761
- [Background] Neuringer M, Sandstrom MM, Johnson EJ, Snodderly DM. Nutritional manipulation of primate retinas, I: effects of lutein or zeaxanthin supplements on serum and macular pigment in xanthophyll-free rhesus monkeys. Invest Ophthalmol Vis Sci. 2004 Sep;45(9):3234-43. doi: 10.1167/iovs.02-1243. PMID 15326146
- [Background] Akbaraly NT, Faure H, Gourlet V, Favier A, Berr C. Plasma carotenoid levels and cognitive performance in an elderly population: results of the EVA Study. J Gerontol A Biol Sci Med Sci. 2007 Mar;62(3):308-16. doi: 10.1093/gerona/62.3.308. PMID 17389729
- [Background] Thomson LR, Toyoda Y, Langner A, Delori FC, Garnett KM, Craft N, Nichols CR, Cheng KM, Dorey CK. Elevated retinal zeaxanthin and prevention of light-induced photoreceptor cell death in quail. Invest Ophthalmol Vis Sci. 2002 Nov;43(11):3538-49. PMID 12407166
- [Derived] Evans JR, Lawrenson JG. Antioxidant vitamin and mineral supplements for slowing the progression of age-related macular degeneration. Cochrane Database Syst Rev. 2023 Sep 13;9(9):CD000254. doi: 10.1002/14651858.CD000254.pub5. PMID 37702300

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were patients in the Ophthalmology/Optometry Clinic North Chicago DVA Medical Center (now the James A. Lovell Federal Health Center)with early and moderate AMD retinopathy up to, but not including,high risk NEI AREDS retinopathy.
Pre-assignment Details: No enrolled participant was excluded before assignment to groups. Patients were asked to continue with their normal diet and were asked not to take any dietary supplement containing lutein (or zeaxanthin) beyond the 250 ug (1/4mg) commonly found in pabulum Centrum® type vitamins.
Groups:
- Lutein: Lutein 9 mg per day
- Lutein Zeaxanthin: 3R 3'R Zeaxanthin 8 mg, Lutein 8 mg per day during 12 months
Period: Overall Study
Arm/Group | Lutein | Lutein Zeaxanthin | Zeaxanthin
Started | 10 | 25 | 25
4 Months | 9 | 24 | 23
8 Months | 9 | 22 | 21
12 Months | 9 | 21 | 21
Completed | 9 | 21 | 21
Not Completed | 1 | 4 | 4
Not completed — Withdrawal by Subject | 0 | 3 | 4
Not completed — Death | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lutein | Lutein Zeaxanthin | Zeaxanthin | Total
Number analyzed (Participants) | 10 | 25 | 25 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 4 | 12
  >=65 years | 7 | 20 | 21 | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 73.9 (9) | 75.8 (9) | 74.4 (11) | 74.9 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 9 | 24 | 24 | 57
Macular Pigment Optical Density [Mean (Standard Deviation); unit: Density units of macular pigment] — Foveal 1 degree estimated central macular pigment density evaluated with the QuantifEye (ZeaVision, Inc., Chesterfield, Missouri),a modified heterochromic flicker photometer (HFP). The MPOD value is derived by taking the logarithm of the ratio between blue and green luminance measured centrally and peripherally. MPOD varies widely between individuals. Low MPOD is 0 - 0.20 density units (du), normal MPOD is 0.20 - 0.50 du and high MPOD is any value above 0.50 du.
  Density units of macular pigment | 0.37 (0.05) | 0.29 (0.06) | 0.35 (0.04) | 0.33 (0.05)
Early Treatment Diabetic Retinopathy Study distance visual acuity [Mean (Standard Deviation); unit: units on a scale] — Black and 10% contrast near reading visual acuity was assessed with a Colenbrander Mixed Contrast Reading Card with LogMAR letters (#4031, Precision Vision, LaSalle, Illinois). We determined single letter acuity on an ordinal VAS (Visual Acuity Scale). The largest letters were 0.05 LogMAR with a VAS = 35 while the most difficult smallest letters were LogMar 1.25 or VAS 105. The test card was held at 40 cm with best monocular refraction, and both low and high contrast letter acuity were assessed.
  units on a scale | 93.3 (8) | 86.8 (12) | 88.3 (10) | 88.7 (13)
Glare Recovery [Mean (Standard Deviation); unit: Seconds] — Photostress glare recovery test involves exposing an individual eye to intense light, or retinal bleach, for a set duration of time and measuring the time taken for visual acuity to recover to a predetermined level. (Margrain 2002) Glare photo-stress recovery (in seconds) following 30 seconds of continuous retinal bleach, was assessed using 2 line supra-threshold low contrast randomly presented Landolt Cs using the KOWA AS14B Night Vision Tester (KOWA Optimed, Tokyo, Japan).
  Seconds | 52.9 (16) | 35.6 (6) | 26.7 (5) | 34.1 (30)
Contrast Sensitivity Function Photopic Distance [Mean (Standard Deviation); unit: units on a scale] — Distance photopic contrast sensitivity function (CSF) at 5 spatial frequencies (1.5, 3, 6, 12 & 20 cc/deg) was determined with the Functional Vision Analyzer® (Stereo Optical Co, Inc, Chicago, IL). Contrast sensitivity readings are shown as a curve. Visual acuity is plotted along the horizontal axis and contrast sensitivity along the vertical axis. Among the normally sighted people, both visual acuity and contrast sensitivity have a wide range of variation.Low population CSF is 0-200 units; normal population CSF is 200-300 units and suprathreshold CSF is 300+ units.
  units on a scale | 212 (34) | 204 (30) | 201 (22) | 204 (125)
Shape Discrimination [Mean (Standard Deviation); unit: % modulation] — We determined the target deformation detection thresholds, or amplitude of the minimum detectable distortion of a 1 degree foveal circular target. The peak spatial frequency of RF (radial frequency) patterns was 5 cyc/deg; the radial modulation frequency was 8 cyc/360°; mean radii were 0.5°, 1°, 2.0°, or 2.5°; and stimulus contrast was 80%. The highest % modulation score possible is 0.13 while the easiest (lowest score) was 10% modulation.
  % modulation | 0.7 (0.2) | 0.7 (0.1) | 1 (0.2) | 0.8 (0.8)
6.5 degrees Tritan threshold [Mean (Standard Deviation); unit: (dB)] — The ChromaTest© is a computerized psychophysical test of protan and tritan color thresholds against age-corrected data. The computer finds the endpoint of the test by a Modified Binary Search method; if response is correct, on the next presentation the color difference between letter and background is halved. If response is incorrect, the color -contrast is doubled. Incorrect responses prolong the test, but do not influence the final threshold. This method of determining thresholds leads to finite steps which reach a plateau at the color contrast sensitivity threshold.
  (dB) | 4.9 (4) | 8.6 (12) | 6 (9) | 6.9 (10)
100% Kinetic Field [Mean (Standard Deviation); unit: Units on a scale (0 to 6000)] — Scotomas within the central 20 degree central macula visual field sensitivity were assessed at 5 contrast levels (20, 40, 60, 80, and full contrast). A yellow wavelength stimulus avoided confounding by the lens. Subjects outline the boundaries of their scotoma(s) on an area-integrating and recording touch flat- screen RGB monitor displaying a central fixation point and movable horizontal/vertical raster lines. The computer calculates summed area of the scotoma(s) with arbitrary scaling from 6000 (dense scotoma) to 0 relative units (absence of scotoma).
  Units on a scale (0 to 6000) | 5514 (2074) | 1717 (765) | 2649 (750) | 2738 (4471)

OUTCOME MEASURES:

1. Primary Outcome: Macular Pigment Optical Density
Description: Replicate measures of foveal 1 degree estimated central MPOD were evaluated with the Quantify® MPS 9000 macular pigment screener, a modified heterochromic flicker photometer (HFP). It employs alternating blue and green flickering LED's and fixation on a 1 degree target, so that a representative measurement at 0.5 degree off center from the fovea is calculated. The method has good repeatability (r = 0.97) and the data are comparable with an objective optical method based on retinal reflectometry (r = 0.78).
Time Frame: 4 months
Population: All participants in all arms were tested
Measure: Mean (Standard Error); unit: Density units of Macular Pigment (du)
Arm/Group | Lutein | Lutein Zeaxanthin | Zeaxanthin
Number analyzed (Participants) | 9 | 24 | 23
Density units of Macular Pigment (du) | 0.48 (.05) | 0.38 (.06) | 0.42 (.04)

2. Secondary Outcome: SHAPE Discrimination
Description: We determined the target deformation detection thresholds, or amplitude of the minimum detectable distortion of a 1 degree foveal circular target. The peak spatial frequency of RF (radial frequency) patterns was 5 cyc/deg; the radial modulation frequency was 8 cyc/360°; mean radii were 0.5°, 1°, 2.0°, or 2.5°; and stimulus contrast was 80%. The highest % modulation score possible is 0.13 while the easiest (lowest score) was 10% modulation.
Time Frame: 12 months
Population: Eyes of all participants still in the trial were measured
Measure: Mean (Standard Deviation); unit: % modulation
Arm/Group | Lutein | Lutein Zeaxanthin | Zeaxanthin
Number analyzed (Participants) | 9 | 21 | 21
% modulation | 0.5 (.24) | 0.6 (0.25) | 0.6 (.46)

3. Secondary Outcome: Early Treatment Diabetic Retinopathy Study Distance Visual Acuity
Description: Black and 10% contrast near reading visual acuity was assessed with a Colenbrander Mixed Contrast Reading Card with LogMAR letters (#4031, Precision Vision, LaSalle, Illinois). We determined single letter acuity on an ordinal VAS (Visual Acuity Scale). The largest letters were 0.05 LogMAR with a VAS = 35 while the most difficult smallest letters were LogMar 1.25 or VAS 105. The test card was held at 40 cm with best monocular refraction, and both low and high contrast letter acuity were assessed.
Time Frame: 12 months
Population: Eyes of all patients still in the trial were measured
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lutein | Lutein Zeaxanthin | Zeaxanthin
Number analyzed (Participants) | 9 | 21 | 21
units on a scale | 98.9 (5.7) | 92.8 (5.9) | 96.8 (8.35)

4. Secondary Outcome: Glare Recovery
Description: Photostress glare recovery test involves exposing an individual eye to intense light, or retinal bleach, for a set duration of time and measuring the time taken for visual acuity to recover to a predetermined level. Glare photo-stress recovery (in seconds) following 30 seconds of continuous retinal bleach, was assessed using 2 line supra-threshold low contrast randomly presented Landolt Cs using the KOWA AS14B Night Vision Tester (KOWA Optimed, Tokyo, Japan).
Time Frame: 12 Months
Population: Eyes of all patients still in the trial were measured
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Lutein | Lutein Zeaxanthin | Zeaxanthin
Number analyzed (Participants) | 9 | 21 | 21
Seconds | 25.2 (28.5) | 14.85 (22) | 16.65 (10.25)

5. Secondary Outcome: Contrast Sensitivity Function Photopic Distance
Description: Distance photopic contrast sensitivity function (CSF) at 5 spatial frequencies (1.5, 3, 6, 12 & 20 cc/deg) was determined with the Functional Vision Analyzer® (Stereo Optical Co, Inc, Chicago, IL). Contrast sensitivity readings are shown as a curve. Visual acuity is plotted along the horizontal axis and contrast sensitivity along the vertical axis. Among the normally sighted people, both visual acuity and contrast sensitivity have a wide range of variation.Low population CSF is 0-200 units; normal population CSF is 200-300 units and suprathreshold CSF is 300+ units.
Time Frame: 12 Months
Population: Eyes of all patients still in the trial were measured
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lutein | Lutein Zeaxanthin | Zeaxanthin
Number analyzed (Participants) | 9 | 21 | 21
units on a scale | 310.5 (33.8) | 247.1 (35) | 254.7 (35.2)

6. Secondary Outcome: 6.5 Degrees Tritan Threshold
Description: The ChromaTest© is a computerized psychophysical test of protan and tritan color thresholds against age-corrected data. The computer finds the endpoint of the test by a Modified Binary Search method; if response is correct, on the next presentation the color difference between letter and background is halved. If response is incorrect, the color -contrast is doubled. Incorrect responses prolong the test, but do not influence the final threshold. This method of determining thresholds leads to finite steps which reach a plateau at the color contrast sensitivity threshold.
Time Frame: 12 months
Population: Eyes of all patients still in the trial were measured
Measure: Mean (Standard Error); unit: dB
Arm/Group | Lutein | Lutein Zeaxanthin | Zeaxanthin
Number analyzed (Participants) | 9 | 21 | 21
dB | 4.46 (1.08) | 8.37 (1.39) | 3.45 (1.09)

7. Secondary Outcome: 100% Kinetic Field
Description: Scotomas within the central 20 degree central macula visual field sensitivity was assessed at 5 contrast levels (20, 40, 60, 80, and full contrast). A yellow wavelength stimulus avoided confounding by the lens. Subjects outlined the boundaries of their scotoma(s) on an area-integrating and recording touch flat- screen RGB monitor displaying a central fixation point and movable horizontal/vertical raster lines. The computer calculated summed area of the scotoma(s) with arbitrary scaling from 6000 (dense scotoma) to 0 relative units (absence of scotoma).
Time Frame: 12 Months
Population: Eyes of all patients still in the trial were measured
Measure: Mean (Standard Error); unit: Units on a scale (0 to 6000)
Arm/Group | Lutein | Lutein Zeaxanthin | Zeaxanthin
Number analyzed (Participants) | 9 | 21 | 21
Units on a scale (0 to 6000) | 2704 (1745) | 2207 (210) | 1129 (650)

8. Primary Outcome: Macular Pigment Optical Density
Description: as for outcome 1
Time Frame: 8 months
Population: All participants in all arms were tested
Measure: Mean (Standard Error); unit: Density units of Macular Pigment (du)
Arm/Group | Lutein | Lutein Zeaxanthin | Zeaxanthin
Number analyzed (Participants) | 9 | 22 | 21
Density units of Macular Pigment (du) | 0.48 (0.05) | 0.44 (0.06) | 0.46 (0.04)

9. Primary Outcome: Macular Pigment Optical Density
Description: Replicate measures of foveal 1 degree estimated central MPOD were evaluated with the Quantify® MPS 9000 macular pigment screener, a modified heterochromic flicker photometer (HFP). It employs alternating blue and green flickering light emitting diodes and fixation on a 1 degree target, so that a representative measurement at 0.5 degree off center from the fovea is calculated.
Time Frame: 12 months
Population: All participants in all arms were tested
Measure: Mean (Standard Error); unit: Density units of Macular Pigment (du)
Arm/Group | Lutein | Lutein Zeaxanthin | Zeaxanthin
Number analyzed (Participants) | 9 | 21 | 21
Density units of Macular Pigment (du) | 0.54 (0.05) | 0.52 (0.06) | 0.48 (0.04)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Lutein and Zeaxanthin have been used as ingredients in dietary supplements since 1994. No adverse report has ever been filed
Arm/Group | Lutein | Lutein Zeaxanthin | Zeaxanthin
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/10 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No